CLINICAL TRIAL: NCT06095544
Title: A Clinical Study on the Application of Enhanced Recovery After Surgery for Simultaneous Pancreas-kidney Transplantation
Brief Title: Enhanced Recovery After Surgery for SPK Transplantation Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2020-hs-67
Record Dates: First submitted 2023-09-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Transplant Complication; Diabetic Nephropathy; Perioperative/Postoperative Complications
Keywords: enhanced recovery after surgery, SPK transplantation
MeSH Terms: conditions — Diabetic Nephropathies; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled tiral
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): ERAS group was consisted of evidenced-based systematic optimization approaches
  Interventions: Procedure: Enhanced recovery for SPK recipients
- Traditional group (No Intervention): The control group received routine care

INTERVENTIONS:
Procedure: Enhanced recovery for SPK recipients — Pre-operative, perioperative and post-operative were consisted of evidenced-based systematic optimization approaches.
  Arms: ERAS group

SUMMARY:
108 patients underwent elective SPK surgery were randomly divided into ERAS group (E) and routine care group (T). The ERAS group was consisted of evidenced-based systematic optimization approaches, while the control group received routine care.

DETAILED DESCRIPTION:
Primary results: the postoperative length of stay (LoS) and hospitalization costs; second results: post-operative analgesia score (NRS) , the incidence of post-operative nausea and vomiting (PONV) , urinary catheter removal time by 7 days , post-operative gastric tube indwelling time, the incidence of ambulation within 6 days . the dosage of dobutamine using , the dosage of norepinephrine using, and the total amount of fluid and urine volume . MAP and lactate level . Peak systolic velocity (PSV) and (resistance index) RI of grafts were checked between two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were aged 20-62 years
2. Body mass index (BMI) of 18.5-32.9 kg/m2
3. Voluntary participation for elective SPK surgery
4. ERSD and DN patients waiting for SPK transplantation surgery.

Exclusion Criteria:

1. History of allergy to narcotic drugs
2. cardiopulmonary insufficiency
3. congestive heart failure
4. myasthenia gravis
5. neurological disease
6. mental illness
7. severe liver dysfunction
8. hyperkalaemia
9. malignant hyperthermia
10. unwilling to participate in the study for any reason, or had participated in another study within the 3 months

Ages: 20 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay (LoS) | Record all the period time from the day of admiting to hospital to the day of discharge from hospital(days).
  Record the time for SPK recipients of LoS (days)
Hospital costs (US dollar) | Total costs(dollar) of the patients spended from the day of admiting to hospital to the day of discharge from hospital(days).
  The total cost of treatment for the patients.

SECONDARY OUTCOMES:
Perioperative complications | After the surgery acomplishment(see detail above)：record the NRS within 40hours after the surgery, occurrence rate of the PPCs within 2 weeks after the surgery, ocurrence rate of the ambulation within 6 days after the surgery, etc.
  48 hours post-operative analgesia score (NRS), the incidence of post-operative nausea and vomiting (PONV) , urinary catheter removal time by 7 days , post-operative gastric tube indwelling time, the incidence of ambulation within 6 days

CONTACTS AND LOCATIONS:
Locations (1):
- Second affiliated hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No